CLINICAL TRIAL: NCT06555120
Title: Screening for Familial Hypercholesterolemia in Children
Acronym: HYPERCHOF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2024_843_0045
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hypercholesterolemia, Familial
Keywords: hypercholesterolemia; familial
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hypercholesterolemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: blood sample — A 5-ml blood sample in a dry tube (or 500-µl cone) is taken and sent to the biochemistry laboratory for lipid analysis.

SUMMARY:
Familial hypercholesterolemia is the most common treatable genetic disorder for which a simple, effective treatment is available, with few side effects.

It leads to a significant increase in LDL levels, generally in excess of 1.9g/l, including in children. It is much higher than the values usually found in secondary or polygenic hypercholesterolemia. This condition multiplies the cardiovascular risk in adulthood by a factor of 13, and is responsible for 6,500 early cardiovascular events per year. In the absence of treatment, the state of the arteries of patients with familial hypercholesterolemia, at the age of 40, would be equivalent to that of 80-year-olds.

Currently, the prevalence is estimated at 1 in 300 people in France. However, this prevalence is largely underestimated, as targeted screening is rarely carried out, and it is estimated that only 10% of sufferers are diagnosed in France, and only 5% of affected children are known and treated.

Today, according to the French health authority, the indications for screening children are: a history of an early vascular event in one of the two parents, or familial hypercholesterolemia in a first-degree relative.

However, the World Health Organization and numerous studies recommend extending screening to the general population. Screening all children and teenagers could make it possible to introduce healthy dietary habits at an early stage, to better adapt the choice of contraception in young women, to treat before the first symptoms appear and thus reduce mortality in adulthood by up to 48%, and to screen relatives who have not yet had a cardiovascular event.

In Slovenia, 90% of children have had a lipid panel since 1994, significantly reducing mortality. In the United Kingdom, the lipid check-up, offered as part of a compulsory visit at the age of two, is being rolled out: 90% of families naturally take it up on the recommendation of their doctors.

The treatment of hypercholesterolemia is simple, and relies first and foremost on hygienic dietary rules and treatments such as statins and Liptruzet (a combination of atorvastatin and ezetimibe), treatments that are easily accessible, effective, with few side effects and low cost.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 and 18 years
* Minimum 8-hour fasting
* Parents and children with signed informed consent

Exclusion Criteria:

* Known familial hypercholesterolemia
* Diabetes less than one month old
* Profound hypothyroidism
* Acute nephrotic syndrome
* cancer under treatment

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
prevalence of hypercholesterolemia in children in the general population | at 16 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No